CLINICAL TRIAL: NCT05704023
Title: Effects of a Mobile App on Adherence to Daily Exercise and Recovery After Whiplash Injury - a Randomized Controlled Trial
Brief Title: Effects of a Mobile App on Adherence to Daily Exercise and Recovery After Whiplash Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blaz Barun (Other)
Responsible Party: Sponsor-Investigator, Blaz Barun, Principal Investigator, University of Split, School of Medicine
Organization: University of Split, School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4090457
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Whiplash Injury of Cervical Spine
Keywords: Whiplash; Adherence; Recovery; Mobile app
MeSH Terms: conditions — Whiplash Injuries

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile app (WIapp) group (Experimental): Standard physical therapy program: 2x10 sessions, 5 times a week, 3-week break in between;
  Mobile app with instructions on exercise at home and daily reminder to exercixse
  Interventions: Behavioral: Reminder to exercise
- Control group (No Intervention): Standard physical therapy program: 2x10 sessions, 5 times a week, 3-week break in between, written instructions on exercises at home

INTERVENTIONS:
Behavioral: Reminder to exercise — Exercise support: Daily, at 7 p.m. patients will get a notification with a reminder to exercise. The app includes photographs of exercises, with instructions, that patients can look at and read if they forget which exercises they need to do and how.
  Arms: Mobile app (WIapp) group

SUMMARY:
This study investigates the effect of daily mobile app reminders to exercise in conjunction with standard physical therapy on adherence to exercise and recovery after whiplash injury of the neck. Participants will be divided into two groups, the experimental (Arm A) and control group (Arm B). Both groups will complete a standard physical therapy program under the supervision of a physiotherapist. Both groups will get illustrated home exercise programs and will be advised to continue exercising at home. In addition, the experimental group will receive one daily push notification via a mobile app to perform a daily exercise at home.

DETAILED DESCRIPTION:
Whiplash injury of the neck is the most common injury resulting from a traffic accident. Although most people recover completely, 30 to 50% of them develop chronic neck pain and disability. Also, long sick leaves and lower productivity at work create a burden on the healthcare system.

Conservative treatment includes exercise, physical therapy modalities such as transcutaneous electric nerve stimulation (TENS), and ultrasound therapy. Although conservative treatment is recommended, the evidence of its efficacy remains unclear. Education after the injury can be beneficial in lowering anxiety and pain.

Many studies are investigating the usefulness of mobile apps in various medical conditions. In rehabilitation medicine, apps are used to increase knowledge about different conditions, as a measurement tool, and as an intervention to increase adherence to the prescribed therapy.

After the enrollment in the study, participants will complete the two-part physical therapy program (2x10 sessions, 5times/day, 3-week break in between) under the supervision of a physiotherapist at the outpatient clinic. After completing the program, the participants will get a home exercise program, group A via mobile app, and group B via papers, and will be encouraged to continue exercising at home. Also, group A will download a mobile app, "WIapp," that was developed for this purpose and will receive one daily push notification as a reminder to perform a daily exercise at home.

The investigators hypothesize that daily reminding to exercise via mobile app can increase adherence to prescribed therapy and overall increase recovery.

ELIGIBILITY:
Inclusion Criteria:

* patients who sustained whiplash injury of the neck in a car accident as drivers or co-drivers
* diagnosed with a whiplash injury of the neck by physical and rehabilitation medicine specialist within 3 months
* Neck Disability Index (NDI) score higher than 5 (10%)
* possession of and ability to use a smartphone and a mobile app
* age ≥ 18 years
* signed written informed consent

Exclusion Criteria:

* bone fracture sustained in the accident
* spinal cord injury
* accident in any other type of vehicle other than car
* treatment of malignant disease in the last 5 years
* expected non-compliance (not possible to use a smartphone because of severe mental or physical impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Change in Neck Disability Index from baseline to 6 months after the injury | baseline, 6 months after the injury
  Physical functioning - where values from 0-8% are regarded as no disability, 10-28% mild disability, 30-48% as moderate disability, 50-68% severe disability, and 70-100% complete disability)

SECONDARY OUTCOMES:
Questionnaire assessment of adherence to exercise | 6 months after the injury
  Adherence to exercise - a 4-point Likert scale regarding weekly exercise completion (classified as: ≥5 sessions/week, 2-4 sessions/week, occasional or no sessions)
Questionnaire assessment of perceived recovery | 6-months after the injury
  Perceived recovery - a 3-point Likert scale on perceived recovery (where 1 indicates non-recovery and 3 indicates full recovery)
Change in Visual Analog Scale (VAS) Pain Score from baseline to 6 months after the injury | baseline, 6 months after the injury
  Pain intensity - ranging from 0 = no pain, to 10 = maximum pain
Pain catastrophizing scale | baseline
  Psychological functioning - (score range from 0-50, a score of 30 or more represents clinically significant level of catastropihizing)
Short Form Health Survey 12 | baseline
  Quality of life - With this questionnaire, it is possible to quantitatively compare physical, psychological, and social consequences caused by impaired health. The score for each question is transformed into standard values and placed on the scale from 0 to 100 (the higher the score the better health) and thus get two major dimensions of health: physical (Physical Common Score-PCS)and mental health (Mental Common Score-MCS).
Questionnaire assessment of social functioning | baseline
  A 5-point Likert scale regarding interference of physical or emotional problems with social function (where 1 indicates constant interference and 5 indicates never)
Questionnaire assessment work | baseline, 6 months after the injury
  The assessment of work with a work status information, a work-time loss and 6-point Likert scale (where 1 indicates normal work capability and 6 indicates no working capability9
Pain catastrophizing scale | 6 months after the injury
  Psychological functioning - (score range from 0-50, a score of 30 or more represents clinically significant level of catastropihizing)
Short Form Health Survey 12 | 6 months after the injury
  Quality of life - With this questionnaire, it is possible to quantitatively compare physical, psychological, and social consequences caused by impaired health. The score for each question is transformed into standard values and placed on the scale from 0 to 100 (the higher the score the better health) and thus get two major dimensions of health: physical (Physical Common Score-PCS)and mental health (Mental Common Score-MCS).
Questionnaire assessment of social functioning | 6 months after the injury
  A 5-point Likert scale regarding interference of physical or emotional problems with social function (where 1 indicates constant interference and 5 indicates never)

CONTACTS AND LOCATIONS:
Overall Officials: Aljinović, Study Director — University Hospital of Split
Locations (1):
- University Hospital Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Barun B, Divic Z, Martinovic Kaliterna D, Poljicanin A, Benzon B, Aljinovic J. Mobile App Intervention Increases Adherence to Home Exercise Program After Whiplash Injury-A Randomized Controlled Trial (RCT). Diagnostics (Basel). 2024 Dec 4;14(23):2729. doi: 10.3390/diagnostics14232729. PMID 39682637